CLINICAL TRIAL: NCT01487967
Title: Preference and Goal-Directed Primary Care to Minimize Disparities and Improve Outcomes in ADHD
Brief Title: Preference and Goal Directed Attention Deficit Hyperactivity Disorder Care- Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-008315
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Preferences; Goals; Decision Making
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Families in the intervention arm will receive culturally appropriate educational material, complete the Preference and Goal Instrument at the study start, use the results to inform decision making about ADHD treatment, have their preferences/goals tracked in the electronic health record, and have their progress toward their goals assessed at 3 months and 6 months (approximately).
  Interventions: Other: Preference and Goal Instrument
- Control (No Intervention): Parents will receive education on ADHD and its treatment, and otherwise receive standard care.

INTERVENTIONS:
Other: Preference and Goal Instrument — Families in the intervention arm will receive culturally appropriate educational material, complete the Preference and Goal Instrument at the study start, use the results to inform decision making about ADHD treatment, have their preferences/goals tracked in the electronic health record, and have their progress toward their goals assessed at 3 months and 6 months (approximately).
  Arms: Intervention

SUMMARY:
This pilot intervention study will test the feasibility and acceptability and explore the outcomes of an urban, primary care-based intervention to measure families' preferences and goals for Attention-Deficit/Hyperactivity Disorder (ADHD) treatment and structure clinical care to reach these goals.

DETAILED DESCRIPTION:
The intervention includes provision of enhanced, culturally appropriate education about ADHD and its treatment, completion of a validated preference and goal instrument, use of this instrument in the ADHD treatment decision-making process, and tracking of preferences and goals over time.

ELIGIBILITY:
Inclusion Criteria:

* All interested non-trainee clinicians at study sites
* Parents/legal guardians of children age 6-12, in K-6 grade, diagnosed with ADHD.

Exclusion Criteria:

* child diagnosed with autism or a psychotic disorder
* parents non-English speaking
* parents unable to provide consent
* pediatric residents

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of family recruitment and follow-up | Up to 24 months
  The feasibility of this intervention will be assessed by examining the proportion of families screened that meet enrollment criteria, the proportion meeting enrollment criteria that enroll, and the proportion enrolled that complete each study measure.

SECONDARY OUTCOMES:
Joint Participation in Decision-Making and Partnership | Baseline
  Participation in decision-making, measured by the Observing Patient Involvement (OPTION) scale.
  Patient partnership, measured by the Patient Participation in Care Scale score after the initial visit at which ADHD treatment decisions are made
Treatment Acceptability | Baseline, after 3 months, after 6 months
  Treatment acceptability measured by the Treatment Acceptability Questionnaire, Parent version (TAQ-P).
Parent Engagement | Up to 24 months
  Engagement will be measured by the number of primary care visits and number of primary care phone calls over the course of the study period
Treatment Adherence/Receipt | Up to 24 months
  Treatment adherence/receipt measured by the number of mental health visits, number of medication refills, and length of time taken to reach a stable treatment dose.
Clinical Outcomes | Baseline, after 3 months, after 6 months
  Change in symptom severity, measured by the Vanderbilt scale over time Change in functional impairment, measured by the Columbia Impairment Scale (CIS), over time
Goal Attainment | after 3 months, after 6 months
  Parents will identify goals at the study start, and progress toward meeting those goals will be tracked during the study.
Acceptability of the intervention to parents and clinicians | Up to 24 months
  Satisfaction with the intervention will be assessed by parent and clinician responses to open-ended questions about satisfaction, acceptability and unintended consequences of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No